CLINICAL TRIAL: NCT02448797
Title: Icotinib as Adjuvant Therapy Compared With Standard Chemotherapy in Stage II-IIIA Non-small Cell Lung Cancer With EGFR-mutation: a Randomized, Positive-controlled, Phase 3 Study (EVIDENCE, CCTC-1501)
Brief Title: Icotinib as Adjuvant Therapy Compared With Standard Chemotherapy in Stage II-IIIA NSCLC With EGFR-mutation
Acronym: EVIDENCE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV-61; CCTC-1501 (Other: China Clinical Trial Consortium)
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Last update posted 2021-07-20 (Actual); Status verified 2020-10

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib; Drug Therapy; Vinorelbine; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- icotinib (Experimental): 125 mg three times daily (375 mg per day) orally for two years.
  Interventions: Drug: Icotinib
- standard chemotherapy (Active Comparator): Vinorelbine 25 mg/m^2, intravenously guttae, day 1 and day 8, 21 days/cycle, 4 cycles.
  cisplatin 75 mg/m^2, intravenously guttae, day 1, 21 days/cycle, 4 cycles.
  For adenocarcinoma: pemetrexed (500 mg/m^2, day 1)/cisplatin (75 mg/m^2, day 1) for 4 cycles.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Icotinib — 125 mg three times daily (375 mg per day) orally for two years.
  Other Names: Conmana
  Arms: icotinib
Drug: Chemotherapy — Vinorelbine 25 mg/m^2, intravenously guttae, day 1 and day 8, 21 days/cycle, 4 cycles, cisplatin 75 mg/m^2, intravenously guttae, day 1, 21 days/cycle, 4 cycles. For adenocarcinoma: pemetrexed (500 mg/m^2, day 1)/cisplatin (75 mg/m^2, day 1) for 4 cycles.
  Other Names: Navelbine; ALIMTA
  Arms: standard chemotherapy

SUMMARY:
Adjuvant therapy has been proved effective in treating earlier stage or less advanced non-small-cell lung cancer. This study is designed to evaluate the efficacy of icotinib as adjuvant therapy in treating stage II-IIIA non-small cell lung cancer patients with EGFR mutation. The primary endpoint is disease-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed non-small cell lung cancer after surgical resection
* Stage II-IIIA disease according to 7th edition of TNM staging
* Positive EGFR gene mutation (19/21)
* ECOG 0-1
* At least 1-year life expectancy
* Adequate organ function

Exclusion Criteria:

* Previous systemic anti-tumor therapy, including chemotherapy or targeted therapy(Including but not limited to monoclonal antibodies, small molecule tyrosine kinase inhibitor, etc
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
* Pneumonectomy of right lung
* Any unresolved chronic toxicity from previous anticancer therapy
* Allergic to study drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2015-06-08 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 48 months
  the time from the date of randomization to the first observation of tumor recurrence, metastasis (based on imaging ) or death

SECONDARY OUTCOMES:
overall survival | 60 months
  The time from the date of randomization to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, MD, Study Chair — Shanghai Pulmonary Hospital, Shanghai, China; Jianxing He, MD, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (8):
- China (8):
  - 307 Hospital of PLA, Beijing, Beijing Municipality
  - Fujian Provincal Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital Of Guangzhou Medical Collage, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Medical School of Zhejiang University, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Occhipinti M, Imbimbo M, Ferrara R, Simeon V, Fiscon G, Marchal C, Skoetz N, Viscardi G. Adjuvant epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors (TKIs) for the treatment of people with resected stage I to III non-small-cell lung cancer and EGFR mutation. Cochrane Database Syst Rev. 2025 May 27;5(5):CD015140. doi: 10.1002/14651858.CD015140.pub2. PMID 40421698
- [Derived] He J, Su C, Liang W, Xu S, Wu L, Fu X, Zhang X, Ge D, Chen Q, Mao W, Xu L, Chen C, Hu B, Shao G, Hu J, Zhao J, Liu X, Liu Z, Wang Z, Xiao Z, Gong T, Lin W, Li X, Ye F, Liu Y, Ma H, Huang Y, Zhou J, Wang Z, Fu J, Ding L, Mao L, Zhou C. Icotinib versus chemotherapy as adjuvant treatment for stage II-IIIA EGFR-mutant non-small-cell lung cancer (EVIDENCE): a randomised, open-label, phase 3 trial. Lancet Respir Med. 2021 Sep;9(9):1021-1029. doi: 10.1016/S2213-2600(21)00134-X. Epub 2021 Jul 21. PMID 34280355